CLINICAL TRIAL: NCT03388333
Title: A Single-center Observational Study to Find Biomarkers for the Outcome of Catheter Ablation in Patients With Atrial Fibrillation
Brief Title: Biomarkers in Patients Undergoing Atrial Fibrillation Ablation
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christian Meyer, Prof. Dr. Christian Meyer, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: D4/17-06
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Atrial fibrillation ablation group: Patients undergoing catheter ablation for the treatment of atrial fibrillation.
  Interventions: Procedure: Catheter Ablation
- Electrophysiological study group: Patients undergoing a diagnostic electrophysiological study without ablation.
- Atrial flutter ablation group: Patients undergoing catheter ablation of right atrial flutter at the cavotricuspid isthmus.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation
  Groups: Atrial fibrillation ablation group; Atrial flutter ablation group

SUMMARY:
The investigators aim to find biomarkers to determine the success of pulmonary vein isolation for the treatment of atrial fibrillation.

DETAILED DESCRIPTION:
The investigators perform an observational study in patients undergoing pulmonary vein ablation to treat atrial fibrillation. Additionally, electrophysiological procedures not related to pulmonary vein isolation are also followed. The aim of the study is finding biomarkers that are able to predict short-term outcome of the procedure.The primary endpoint is defined as reoccurrences of atrial fibrillation within the first three months after pulmonary vein isolation.

ELIGIBILITY:
Inclusion Criteria:

* patients with atrial fibrillation scheduled for pulmonary vein isolation with either radiofrequency of cryoballoon
* patients scheduled for an electrophysiological study without ablation
* patients with a catheter ablation at the cavotricuspid isthmus for the treatment of right atrial flutter

Exclusion Criteria:

* patients with concurrent pulmonary vein isolation and ablation of the cavotricuspid isthmus
* Acute myocardial infarction, coronary artery bypass graft surgery or open heart surgery within less than 3 months prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation schedulded for pulmonary vein isolation
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with short term reoccurrences of atrial fibrillation after ablation. | 3 months
  Holter ECGs and ECGs after atrial fibrillation ablation

SECONDARY OUTCOMES:
Change in heart rate after pulmonary vein isolation | 3 days.
  Heart rates are recorded at admission and release from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, Prof. Dr., Principal Investigator — Germany Department of Cardiology - Electrophysiology, University Heart Centre
Locations (1):
- Department of Cardiology - Electrophysiology, University Heart Centre, University Hospital Hamburg-Eppendorf, Hamburg, Germany